CLINICAL TRIAL: NCT06605664
Title: Hyperpolarized 13C-MRI, Metabolomics, and Radiomics for Immune Response Prediction in Patients With Hepatocellular Carcinoma Undergoing Radiotherapy, Atezolizumab, and Bevacizumab
Brief Title: Hyperpolarized 13C-MRI in Patients With Hepatocellular Carcinoma Undergoing Radiotherapy, Atezolizumab, and Bevacizumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Cheng-En Hsieh, Attending Physician, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2401190005
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hyperpolarized 13C-MRI; HCC; Radiotherapy; Metabolomics; Atezolizumab; Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Single arm of hyperpolarized 13C pyruvate MRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperpolarized 13C pyruvate MRI (Experimental): Hyperpolarized 13C pyruvate MRI before and 2-5 weeks after radiotherapy combined with atezolizumab and bevacizumab
  Interventions: Diagnostic Test: Hyperpolarized 13C pyruvate MRI

INTERVENTIONS:
Diagnostic Test: Hyperpolarized 13C pyruvate MRI — The subject enrolled in this trial will receive DNP-MRI scanning for two times through hyperpolarized [1-13C]pyruvate injection (~250 mM, 0.43 mL/Kg) before and 2-5 weeks after radiotherapy.

SUMMARY:
Increased pyruvate-to-lactate conversion is a hallmark of HCC metabolism. In parallel, activation of pro-inflammatory immune cells triggers a metabolic switch towards anaerobic glycolysis. Hyperpolarized carbon-13 (13C) pyruvate MRI is a state-of-the-art non-invasive imaging method that offers real-time insights into tissue metabolism. Recent studies have demonstrated its promising potential in predicting responses to radiotherapy and immunotherapy in solid tumors, given the significance of pyruvate as a downstream metabolite in glycolysis. However, its application in assessing treatment response in hepatocellular carcinoma (HCC) patients remains unclear. The establishment of quantitative imaging biomarkers for predicting responses to radio-immunotherapy is an unmet need in the management of HCC patients.

While radiotherapy (RT) effectively controls localized tumors through the induction of unrepairable DNA double-stranded breaks (DSBs) and cell death, its therapeutic efficacy on distal, non-irradiated tumor cells is limited, with out-of-field recurrence being a common pattern of failure in HCC patients treated with high-dose irradiation. Atezolizumab (anti-programmed death-ligand 1; anti-PD-L1) in conjunction with bevacizumab (anti-vascular endothelial growth factor; anti-VEGF) has recently emerged as the standard first-line systemic treatment for unresectable hepatocellular carcinoma (HCC). Despite an objective response rate (ORR) of only 27%, the majority of patients succumb to HCC progression and liver failure. Our preclinical study (Hsieh et al., Science Immunology 2022) uncovered that RT, when combined with PD-L1/PD-1 blockade, induces immunogenic cell death and tumor antigen cross-presentation in antigen-presenting cells, enhancing systemic antitumor T cell responses in murine tumor models. Recent retrospective cohorts suggest that RT targeting all hepatic tumors combined with PD-L1/programmed death-1 (PD-1) blockade is associated with an improved ORR and median progression-free survival (PFS) in patients with unresectable HCC, demonstrating a favorable safety profile. The synergistic antitumor effects of this combination therapy with RT, atezolizumab, and bevacizumab have led to its increasing adoption in routine clinical practice.

This phase II non-randomized trial aims to prospectively investigate the predictive value of hyperpolarized 13C-MRI, along with comprehensive metabolomics and radiomics analyses, for immune response assessment including tumor control outcomes and toxicity in patients with HCC undergoing radiotherapy, atezolizumab, and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have diagnosis of HCC that is deemed unsuitable for surgical resection or transplant and will undergo radiotherapy, atezolizumab, and bevacizumab. Participants may have multiple lesions with a total maximal tumor dimension of < 20 cm, and no one lesion > 15 cm. Diagnosis should be confirmed by at least 1 criteria listed below:

   * Histologically or cytologically proven diagnosis of HCC.
   * Typical arterial enhancement and delayed washout on multiphasic CT or MRI.
2. Age ≥18 years at the time of signing informed consent document.
3. ECOG performance status 0-1.
4. Barcelona Clinic Liver Cancer (BCLC) stages Intermediate (B) or Advanced (C).
5. Child-Pugh score 5-6 liver function within 28 days of study registration.
6. Documented virology status of hepatitis B virus (HBV), as confirmed by screening HBV serology test.
7. Documented virology status of hepatitis C virus (HCV), as confirmed by screening HCV serology test.
8. Ability to understand and the willingness to sign a written informed consent document
9. Adequate bone marrow, liver, and renal function within 4 weeks before study registration

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,000/mm3
   * Platelet count ≥ 50,000/μL
   * Total bilirubin < 2.5 mg/dL
   * Serum albumin >2.8 g/dL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN)
   * Prothrombin time ≤ 6 seconds prolonged
   * Serum creatinine ≤ 1.5 mg/dL
10. The medical team, experienced in liver cancer treatment, has evaluated and confirmed that the benefits outweigh the risks for participants receiving proton or photon radiation therapy combined with atezolizumab and bevacizumab.

Exclusion Criteria:

1. Prior invasive malignancy unless disease free for a minimum of 2 years
2. Prior radiotherapy to the region of the liver that would result in overlap of radiation therapy fields
3. Prior selective internal radiotherapy/hepatic arterial yttrium therapy, at any time
4. Untreated active hepatitis B or hepatitis C
5. Moderate to severe or intractable ascites
6. Presence of distant metastases
7. Untreated or incomplete treated esophageal or gastric varices
8. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
   * Myocardial infarction within the last 6 months prior to study entry
   * Acute bacterial or fungal infection requiring intravenous antibiotics within 28 days prior to study entry
   * A bleeding episode within 6 months prior to study entry due to any cause.
   * Thrombolytic therapy within 28 days prior to study entry.
   * Known bleeding or clotting disorder.
   * Uncontrolled psychotic disorder
9. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
10. Prior solid organ transplantation.
11. Prior or active autoimmune disease (AID) including autoimmune hepatitis, inflammatory bowel disease, myasthenia gravis, systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, and multiple sclerosis.
12. Prior or active thrombotic or bleeding disorders, hemoptysis, cerebral vascular accident, significant cardiac disease (ischemic or congestive heart failure), or gastrointestinal perforation.
13. Inability to treat all sites of disease by proton radiotherapy (such as extrahepatic metastases or massive liver tumors whereby the liver constraints cannot be met for covering all sites of liver tumors using radiotherapy.)
14. Known HIV infection.
15. Conditions not suitable for magnetic resonance imaging (MRI) include the presence of strongly magnetic arterial clips in the brain, cardiac pacemakers, cochlear implants, and claustrophobia.
16. Concurrent medical conditions that may impact patients during MRI examination include active infections, symptomatic congestive heart failure, uncontrollable angina, arrhythmias, mental disorders, difficulty breathing, or diarrhea.
17. An endoscopy report within the past six months indicates a high risk for upper gastrointestinal bleeding, and the patient has not received complete treatment for its prevention.
18. Individuals who are allergic to hyperpolarized 13C pyruvate, atezolizumab, bevacizumab, or any ingredients contained in these medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic Nuclear Polarization (DNP) | 4 months
  Dynamic Nuclear Polarization (DNP) conversion flux (pyruvate-to-lactate conversion rate [Kpl] and area under the curve [AUC]) before radiotherapy combined with atezolizumab and bevacizumab
Dynamic Nuclear Polarization (DNP) | 4 month
  Dynamic Nuclear Polarization (DNP) conversion flux (pyruvate-to-lactate conversion rate [Kpl] and area under the curve [AUC]) 2-5 weeks after radiotherapy combined with atezolizumab and bevacizumab

SECONDARY OUTCOMES:
Progression free survival (PFS) by RECIST1.1 | 12 months
  PFS is defined as the time from signing the informed consent to the first occurrence of disease progression or death from any cause (whichever occurs first) according to RECIST1.1
Local control (LC) by RECIST1.1 | 12 months
  LC is defined as the time from signing the informed consent to the first occurrence of disease progression in the irradiated field according to RECIST1.1
Time to progression (TTP) by RECIST1.1 | 12 months
  TTP is defined as the time from signing the informed consent to the first occurrence of disease progression according to RECIST1.1
Overall Response Rate (ORR) by RECIST1.1 | 12 months
  ORR is defined as a complete or partial response according to RECIST1.1
Overall survival (OS) | 12 months
  OS is defined as the time from signing the informed consent to death from any cause.
Incidence and severity of adverse events | 12 months
  Adverse events will be graded using CTCAE v5

OTHER OUTCOMES:
Change in myeloid-derived suppressor cell (MDSC) level in peripheral blood | 4 months
  We will measure the level of Lin- HLA-DR- CD11b+ MDSCs in peripheral blood using flow cytometry before and 2-5 weeks after radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of individual participant data (IPD) requires IRB approval.